CLINICAL TRIAL: NCT01635062
Title: Evaluating Hormonal Mechanisms for Vitamin D Receptor Agonist Therapy in Diabetes: The VALIDATE-D Study
Brief Title: The VALIDATE-D Study
Acronym: VALIDATE-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Anand Vaidya, Assistant Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2012P000905
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- calcitriol (Experimental): Subjects will receive calcitriol (titrated up to 0.75 mcg daily) for 3 weeks.
  Interventions: Drug: Calcitriol
- placebo (Placebo Comparator): Subjects will receive placebo for 3 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcitriol — Subjects will receive calcitriol (up to 0.75 mcg daily) for 3 weeks.
  Other Names: 1,25-dihydroxyvitamin D3
  Arms: calcitriol
Drug: Placebo — Subjects will receive placebo for 3 weeks.
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate whether vitamin D receptor agonist therapy lowers renin-angiotensin system activity.

DETAILED DESCRIPTION:
This study aims to evaluate whether vitamin D receptor agonist therapy (calcitriol) in diabetes lowers renin-angiotensin system (RAS) activity in a manner similar to an ACE inhibitor. This is a physiology study, focused on evaluating hormonal changes in the circulating and tissue RAS when compared to placebo.

Subjects with type 2 diabetes and obesity and normal kidney function will undergo evaluation of their circulating and renal-vascular RAS activity and urinary protein at baseline, after withdrawing interfering medications, while on a controlled electrolyte diet, and in controlled posture settings. They will then randomly receive a study medication (calcitriol or placebo) for 3 weeks followed by a re-assessment of their RAS parameters. The main outcomes that will be evaluated following calcitriol/placebo include measures of the circulating renin activity (primary), as well as measures of the renal-vascular RAS (renal plasma flow) and urine protein (secondary)

The primary outcome is the change in the plasma renin activity when sodium restricted, before and after intervention. Secondary outcomes include the change in renal plasma flow and urine protein when sodium loaded, before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Type-Two Diabetes (treated with diet alone, with oral hypoglycemic agents, or with a single injection of basal insulin daily)
2. Normal blood pressure, or Mild (Stage 1) Hypertension that is either untreated, or adequately treated with a single anti-hypertensive drug.
3. Age >18 years and <70 years
4. Estimated GFR > 60ml/min
5. Normal laboratory values for: Complete blood count, sodium, potassium, glucose, liver enzymes, urinalysis
6. Electrocardiogram without any signs of prior infarction, ventricular conduction abnormality, or supraventricular arrhythmia.

Exclusion Criteria:

1. Chronic Kidney Disease or eGFR<60
2. History of nephrolithiasis (kidney stones)
3. Multiple (more than one) insulin injections daily (since insulin can alter the RAS)
4. Poorly controlled type 2 diabetes (That may require more aggressive therapy) as defined by an HbA1c>8.5%
5. Type 1 diabetes
6. Stage 2 or Stage 3 hypertension or the use of more than 1 antihypertensive drug
7. Chronic inflammatory conditions (such as inflammatory bowel disease or arthritis) that are treated with prescribed doses of NSAIDs by a physician.
8. The use of prescribed doses of potassium supplements.
9. History of liver failure
10. History of parathyroid or granulomatous disorders
11. History of heart failure, cerebrovascular disease or coronary heart disease
12. History of known microvascular complications of diabetes (including retinopathy, neuropathy, nephropathy)
13. Illness requiring overnight hospitalization in the past 6 months
14. Active tobacco or recreational drug use
15. Pregnancy or current breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Vaidya, MD, MMSc, Principal Investigator — Brigham and Women's Hospital, Harvard Medical School
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Brown JM, Secinaro K, Williams JS, Vaidya A. Evaluating hormonal mechanisms of vitamin D receptor agonist therapy in diabetic kidney disease: the VALIDATE-D study. BMC Endocr Disord. 2013 Aug 23;13:33. doi: 10.1186/1472-6823-13-33. PMID 23971740

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the local Boston community
  A total of 41 participants were consented to participate. Subsequently, 13 were found ineligible, 5 withdrew participation, 3 were lost-to follow-up, and 2 were withdrawn for non-compliance with the washout. Therefore, 18 were randomized.
Pre-assignment Details: An anti-hypertensive medication washout was conducted to minimize confounding of the renin-angiotensin system.
  ACE inhibitors, angiotensin-receptor blockers, and mineralocorticoid receptor antagonists, beta blockers, diuretics, and calcium-channel blockers were withdrawn for 2 weeks to 2 months prior to randomization.
Groups:
- Calcitriol: Subjects will receive calcitriol (titrated up to 0.75 mcg daily) for 3 weeks.
  Subjects have their renin-angiotensin system, renal plasma flow, and urine protein assessed at baseline while sodium restricted and sodium loaded. They will then be randomized to receive calcitriol (up to 0.75 mcg daily) or placebo for 3 weeks, and repeat assessments again while sodium restricted and sodium loaded.
- Placebo: Subjects will receive placebo for 3 weeks.
  Subjects have their renin-angiotensin system, renal plasma flow, and urine protein assessed at baseline while sodium restricted and sodium loaded. They will then be randomized to receive calcitriol (up to 0.75 mcg daily) or placebo for 3 weeks, and repeat assessments again while sodium restricted and sodium loaded.
Period: Overall Study
Arm/Group | Calcitriol | Placebo
Started | 9 | 9
Sodium Restriction Baseline Visit (The first study visit was a pre-randomization assessment while sodium restricted (Baseline)) | 9 | 9
Sodium Loading Baseline Visit (The second study visit was a pre-randomization assessment while sodium loaded (Baseline)) | 9 | 9
Post-randomization Sodium Restriction (This visit was an assessment while sodium restricted and following 3 weeks of study medication) | 9 | 9
Post-Randomization Sodium Loaded (This visit was an assessment while sodium loaded and following 3 weeks of study medication) | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcitriol | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (10.4) | 50.7 (5.0) | 50.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 7 | 4 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: The Change in Circulating RAS Activity After Calcitriol/Placebo Therapy
Description: The below results represent the change in Plasma Renin Activity.
Time Frame: baseline and 2 weeks following calcitriol/placebo therapy
Measure: Median (Inter-Quartile Range); unit: ng/mL/h
Groups:
- Calcitriol; Placebo: Subjects have their plasma renin activity assessed at baseline while sodium restricted, and again after 2 weeks of randomized therapy with calcitriol (up to 0.75 mcg daily) or placebo.
Arm/Group | Calcitriol | Placebo
Number analyzed (Participants) | 9 | 9
ng/mL/h | 0 [-1.3 to 0.3] | -1.3 [-3.6 to -0.3]
Statistical Analysis 1: Comparison: Calcitriol vs Placebo; The hypothesis was that calcitriol therapy would lower plasma renin activity (PRA), when sodium restricted, when compared to placebo; Test type: Superiority or Other; p = 0.69, ANOVA; Median Difference (Final Values) = 1.3

2. Secondary Outcome: Change in Renal Plasma Flow After Calcitriol/Placebo Therapy
Description: Subjects had their renal plasma flow assessed at baseline while sodium loaded, and again after 3 weeks of randomized therapy with either calcitriol (up to 0.75 mcg daily) or placebo.
Time Frame: baseline and 3 weeks following calcitriol/placebo therapy
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Groups:
- Calcitriol; Placebo: Subjects have their renal plasma flow assessed at baseline while sodium loaded. They will then be randomized to receive calcitriol (up to 0.75 mcg daily) or placebo for 3 weeks, and repeat renal plasma flow assessments again while sodium loaded.
Arm/Group | Calcitriol | Placebo
Number analyzed (Participants) | 9 | 9
mL/min/1.73m2 | -16.4 (180.5) | -0.6 (142.2)
Statistical Analysis 1: Comparison: Calcitriol vs Placebo; The hypothesis was that calcitriol therapy would raise renal plasma flow, when sodium loaded, when compared to placebo; Test type: Superiority or Other; p = 0.89, ANOVA; Mean Difference (Final Values) = 15.8

3. Secondary Outcome: Change in Urine Protein After Calcitriol/Placebo Therapy
Description: Subjects have their urine protein assessed at baseline while sodium loaded and again 3 weeks after randomized therapy with calcitriol or placebo.
Time Frame: baseline and 3 weeks following calcitriol/placebo therapy
Measure: Mean (Standard Deviation); unit: mg/24h
Groups:
- Calcitriol; Placebo: Subjects have their urine protein assessed at baseline while sodium sodium loaded and again following 3 weeks of randomization to calcitriol (up to 0.75 mcg daily) or placebo.
Arm/Group | Calcitriol | Placebo
Number analyzed (Participants) | 9 | 9
mg/24h | 21.1 (95.7) | 8.1 (51.0)
Statistical Analysis 1: Comparison: Calcitriol vs Placebo; The hypothesis was that calcitriol therapy would lower urine protein, when sodium loaded, when compared to placebo; Test type: Superiority or Other; p = 0.80, ANOVA; Mean Difference (Final Values) = 13.0

ADVERSE EVENTS:
Time Frame: They were collected for the duration of the study (~4 months)
Arm/Group | Calcitriol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

LIMITATIONS AND CAVEATS:
This was a small physiological study, not a treatment study or a typical Phase 1-4 study. The objective was to investigate the mechanistic link between vitamin D receptor agonist therapy and the renin-angiotensin system.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No